CLINICAL TRIAL: NCT05860127
Title: Cognitive Stimulation Therapy for Dementia: A Two-Armed Pragmatic Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Amherst (Other)
Collaborators: Yale University (Other); UConn Health (Other); National Institute on Aging (NIA) (NIH); University of Maryland, Baltimore (Other)
Responsible Party: Principal Investigator, Michael Lepore, Professor, University of Massachusetts, Amherst
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00054748; 5U54AG063546-04 (NIH)
Record Dates: First submitted 2023-02-14; First posted 2023-05-16 (Actual); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Dementia; Cognitive Impairment, Mild; Dementia, Vascular; Dementia, Mixed; Dementia With Lewy Bodies; Dementia Frontal; Dementia Moderate; Dementia of Alzheimer Type; Dementia, Mild
MeSH Terms: conditions — Dementia; Cognitive Dysfunction; Dementia, Vascular; Mixed Dementias; Lewy Body Disease; Lymphoma, Follicular | interventions — Referral and Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Referral for Cognitive Stimulation Therapy (Active Comparator): This group will receive a referral from their physician for CST treatment
  Interventions: Behavioral: Referral for Cognitive Stimulation Therapy
- Standard of Care (Placebo Comparator): This group will receive standard of care and no CST referral.
  Interventions: Other: No change to Standard of Care

INTERVENTIONS:
Behavioral: Referral for Cognitive Stimulation Therapy — Physician will review participant eligibility for CST treatment and offer referral based on clinical judgement
  Arms: Referral for Cognitive Stimulation Therapy
Other: No change to Standard of Care — Participants will not receive referral from a physician. They will continue with standard of care at their site.
  Arms: Standard of Care

SUMMARY:
Cognitive Stimulation Therapy (CST) is an evidence-based non-pharmacological group therapy shown to benefit people with mild to moderate dementia. Despite increasing availability of CST worldwide, access remains limited in the United States. This pilot pragmatic trial will embed CST referral into the standard care protocol of health care settings that serve people living with dementia in the state of Connecticut, and evaluate online delivery of CST known as virtual CST (V-CST), and assess the acceptability of V-CST to people living with dementia.

The study design is a two-armed randomized embedded pragmatic clinical trial (ePCT). The trial aims to determine if cognitive decline is experienced less commonly among V-CST participants than control group members based on three widely used measures of cognition, the Montreal Cognitive Assessment (MoCA), St. Louis University Memory Screen (SLUMS), and Mini Mental State Exam (MMSE).

The study population will be persons with mild to moderate dementia identified by clinicians in standard care. From this population, subject participants will be randomized to intervention and control groups. Patients randomly assigned to the intervention group will be referred by their clinical providers to participate in V-CST, and those who accept the referral will participate in the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Mild Cognitive Impairment or Mild to Moderate Dementia
* MoCA score of 10 to 26 OR SLUMS score of 10 to 26 OR MMSE score between 13 and 24 recorded as present < 24 months before the record review
* English-speaking
* Visit scheduled to include cognitive screening 6 to 12 months after record review.

Exclusion Criteria:

* Auditory or visual impairment, combative behaviors, or other clinician-assessed condition that would interfere with group treatment
* No access to online meeting platform
* Patient has specified to HCS not to engage patient in research or to use patient data in research
* Patient has previously participated in V-CST
* Physician determines a caregiver is needed to support V-CST participation, but no caregiver available to assist with technology.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2023-04-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Cognitive decline measured by an increase in Montreal Cognitive Assessment Score from baseline to follow-up | 6 months
  Clinically meaningful cognitive decline will be less common in intervention group than the control group. Clinically meaningful changes will be assessed using one of the following cognitive assessment tools: Montreal Cognitive Assessment (MoCA), Saint Louis University Mental Status (SLUMS) exam, or the Mini-Mental State Examination (MMSE). A 'crosswalk' will be used to convert all cognitive assessment measures to a MoCA score. All participants will start with a baseline MoCA score of 10 to 26 which indicates mild-moderate cognitive impairment. An increase in the baseline MoCA score by 2 points or greater indicates a clinically meaningful decline in cognitive status. Cognitive assessments will be collected at baseline and 6 months follow-up visit after baseline/enrollment. All cognitive assessments will be done by the study physicians. The cognitive assessment collected at baseline will be the cognitive assessment used to assess cognitive impairment at the 6 month follow-up.

SECONDARY OUTCOMES:
Cognitive improvement measured by a decrease in Montreal Cognitive Assessment Score from baseline to follow-up | 6 months
  Clinically meaningful cognitive improvement will be more common in the intervention group than the control group. Clinically meaningful changes will be assessed using one of the following cognitive assessment tools: Montreal Cognitive Assessment (MoCA), Saint Louis University Mental Status (SLUMS) exam, or the Mini-Mental State Examination (MMSE). A 'crosswalk' will be used to convert all cognitive assessment measures to a MoCA score. All participants will start with a baseline MoCA score of 10 to 26 which indicates mild-moderate cognitive impairment. A decrease in the baseline MoCA score by 2 points or greater indicates a clinically meaningful improvement in cognitive status. Cognitive assessments will be collected at baseline and 6 months follow-up visit after baseline/enrollment. All cognitive assessments will be done by the study physicians. The cognitive assessment collected at baseline will be the cognitive assessment used to assess cognitive impairment at the 6 month follow-up.
Referral Acceptance Rate | 1 month
  V-CST referral will be favorably received by participants. V-CST referral will be assessed by referral acceptance rate measured by percentage of people referred for V-CST who accept the referral over the 1-month referral period process. This outcome will be assessed at the end of the referral process.
Participant attendance | 7 weeks
  V-CST treatment will be favorably received by participants. Participant attendance will be measured as the percentage of enrolled participants who attend each V-CST session. V-CST sessions will be conducted over a 7-week period. This outcome will be assessed at the end of the 7th week V-CST session.
Participant Attrition | 7 weeks
  V-CST treatment will be favorably received by participants. Participant attrition will be measured as the percentage of enrolled participants who cease attending V-CST between session 1 and session 14. V-CST sessions will be conducted over a 7-week period. This outcome will be assessed at the end of the 7th week V-CST session.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lepore, PhD, Principal Investigator — University of Massachusetts, Amherst
Locations (2):
- United States (2):
  - UConn Center on Aging, Farmington, Connecticut
  - Yale Memory Clinic, New Haven, Connecticut

IPD SHARING:
Plan to Share IPD: No